CLINICAL TRIAL: NCT04108845
Title: A Single-center, Open, Phase I Clinical Trial to Evaluate Safety of 15-Valent Pneumococcal Conjugate Vaccine in Healthy Volunteers Aged Above 2 Months
Brief Title: Safety Study of 15-Valent Pneumococcal Conjugate Vaccine in Healthy Volunteers Aged Above 2 Months
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Collaborators: Hebei Center for Disease Control and Prevention (Unknown); Laishui Center for Disease Control and Prevention (Unknown); National Institutes for Food and Drug Control, China (Other); Simoon Record Pharma Information Consulting Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201807001
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Pneumonia, Pneumococcal
MeSH Terms: conditions — Pneumonia, Pneumococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Received Vaccine: 15-valent pneumococcal Conjugate Vaccine, 0.5 ml/dose
  Interventions: Biological: 15-Valent Pneumococcal Conjugate Vaccine

INTERVENTIONS:
Biological: 15-Valent Pneumococcal Conjugate Vaccine — 3/1 dose(s) according to age of subjects. Single intramuscular dose contains 0.5ml 15-Valent Pneumococcal Conjugate Vaccine.

SUMMARY:
The purpose of this study is to evaluate safety of 15-Valent Pneumococcal Conjugate Vaccine in healthy volunteers aged above 3 Months.

ELIGIBILITY:
Inclusion Criteria:

* 2 months old (at a minimum of 6 weeks old) and above healthy people.
* Subject or legal representative who consent and has signed written informed consent.
* Subject and parent/guardian who is able to comply with all study procedures and to use thermometer, scale and fill in diary card and contact card as required.
* Subject who didn't vaccinate 13-valent or 7-valent pneumococcal conjugate vaccine.
* Subject who did't immune with any live vaccine within 14 days and inactivated vaccine within 7 days before vaccination.
* Axillary temperature ≤37.0 ℃.

Exclusion Criteria:

* Subject with a history of a prior bacterial culture of an aggressive disease caused by S. pneumoniae.
* Subject with any previous history of severe vaccination or drug allergy, occurrence of fever ≥ 39.0° related to vaccination of biological products for previous vaccination.
* Subject who are allergic to diphtheria toxins.
* Children below 1 year old with abnormal labor（dystocia, instrument midwifery), birth weight <2500g, asphyxia rescue history, nerve organ damage history, and pathological history of yellow plague determined by diagnosis.
* History of allergy，eclampsia, epilepsy,brain trauma,encephalopathy and mental disease or family disease.
* Subject who diagnosis of thrombocytopenia or other history of coagulopathy.
* Known severe congenital malformations, developmental disorders; clinically diagnosed serious chronic diseases: down's syndrome, diabetes, sickle cell anemia or neurological disorders, Guillain Barre syndrome.
* Known or suspected to suffer from: severe cardiovascular disease, liver and kidney disease, malignant tumor, skin disease, serious respiratory system disease, acute infection or chronic disease active period.
* Known or suspected to suffer from immunological abnormalities, including immunosuppressive therapy (radiotherapy, chemotherapy, corticosteroids, antimetabolic drugs, cytotoxicity drugs), HIV infection, etc.
* Received blood products or immunoglobulin within 3 months before enrolling (hepatitis B immunoglobulin was acceptable), or planned to use it during the clinical trial period (before blood samples were collected after immunization).
* Subject who plan to participate in or is in any other clinical trial (vaccines, drugs, medical devices, etc.).
* In pregnancy or lactation or pregnant women.
* ≥18-year-old subject with blood routine, blood chemistry or urinalysis laboratory collection abnormalities.
* Any condition that, in the judgment of investigator, may affect trial assessment.

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events in 30 minutes | 30 minutes after each vaccination
  Occurrence of adverse events in 30 minutes after each vaccination
Solicited adverse events during 7 days | 7 days after each vaccination
  Occurrence of solicited adverse events during a 7-day follow-up period after each vaccination
Unsolicited adverse events during 30 days | 30 days after each vaccination
  Occurrence of unsolicited adverse events during a 30-day follow-up period after each vaccination
SAE | from enrolling to 6 months after all vaccinations
  Occurrence of serious adverse events (SAE) from enrolling to 6 months after all vaccinations
Blood routine of subjects over 18 years old at the fourth day | 4 days after vaccination
  Blood routine test results of subjects over 18 years old at the fourth day after vaccination
Blood biochemistry of subjects over 18 years old at the fourth day | 4 days after vaccination
  Blood biochemistry test results of subjects over 18 years old at the fourth day after vaccination
Urine routine of subjects over 18 years old at the fourth day | 4 days after vaccination
  Urine routine test results of subjects over 18 years old at the fourth day after vaccination

SECONDARY OUTCOMES:
Subjects ratio of vaccine serotype specific pneumococcal IgG antibody concentration ≥ 0.35 ug/ml or 1.0 ug/ml in 2-month-old and 3-month-old subjects | 30 days after immunization
  Subjects ratio of vaccine serotype specific pneumococcal IgG antibody concentration ≥ 0.35 ug/ml or 1.0 ug/ml in 2-month-old and 3-month-old subjects on 30 days after immunization with 15-valent pneumococcal polysaccharide conjugate vaccine
GMC of vaccine serotype specific pneumococcal IgG antibody in 2-month-old and 3-month-old subjects | 30 days after immunization
  Geometric mean concentration (GMC) of vaccine serotype specific pneumococcal IgG antibody in 2-month-old and 3-month-old subjects on 30 days after immunization with 15-valent pneumococcal polysaccharide conjugate vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Du Lin, Master, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Laishui Center for Disease Control and Prevention, Laishui, Hebei, China

IPD SHARING:
Plan to Share IPD: No